CLINICAL TRIAL: NCT02875522
Title: The Effects of Aerobic Exercise Training on Peripheral Vascular, Cardiac and Cerebral Vascular Function in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Effects of Aerobic Exercise Training on Vascular, Cardiac and Cerebral Vascular Function in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H11-02770
Record Dates: First submitted 2016-08-04; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Exercise Training; Flow-Mediated Dilation; Arterial Stiffness; Echocardiography; Cerebrovascular Physiology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Patients with COPD (Experimental): Stable patients with COPD participated in an 8-week (24 session) individualized, non-linear aerobic exercise training program consisting of upper and lower body cycle ergometry.
  Interventions: Other: Individualized, non-linear aerobic exercise training
- Healthy Controls (Active Comparator): Age, sex, BMI and activity matched controls participated in an 8-week (24 session) individualized, non-linear aerobic exercise training program consisting of upper and lower body cycle ergometry.
  Interventions: Other: Individualized, non-linear aerobic exercise training

INTERVENTIONS:
Other: Individualized, non-linear aerobic exercise training — Aerobic exercise performed on lower body stationary ergometer and an upper extremity arm crank. Intensity (50-95% workload maximum) and durations (20-45 min) are fluctuated daily to optimize training stress and adaptation

SUMMARY:
The primary cause of chronic obstructive pulmonary disease is smoking, which can lead to inflammation in the lungs and blood vessels that can lead to secondary problems such as blood vessel disease, high blood pressure and heart disease. Aerobic exercise training has been shown to reduce the risk of heart and brain disease; however, it is currently unknown whether exercise training can have the same affect in patients with COPD. The aim of this study is to investigate how eight weeks of aerobic exercise training improves blood vessel and heart function and brain blood flow in patients with COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a treatable respiratory condition that is only partially reversible. The primary cause of COPD is smoking which leads to airway inflammation and oxidative damage to the lungs, which has been linked to the development and progression of the disease. The inflammation is not isolated to the lungs as patients with COPD also have systemic inflammation that has been linked to a number of cardiovascular comorbidities such as endothelial dysfunction, cardiovascular disease and stroke. Evidence demonstrates that COPD patients have a greater incidence of vascular dysfunction and adverse vascular remodeling, which worsens with disease severity. In fact, patients with COPD are at 35 times greater risk of developing cardiovascular disease and stroke than healthy aged matched individuals. In healthy individuals and a number of chronic conditions, aerobic exercise training is well established to reduce the risk of cardiovascular and cerebrovascular disease. The benefits of exercise are likely through improvements in endothelial function, systemic inflammation, and cardiac and cerebral vascular function. However, whether exercise training can have the same effects in a chronic inflammatory condition like COPD has not been studied. The purpose of this study is to determine the effectiveness of an 8 week aerobic exercise training program in patient's chronic obstructive pulmonary disease as determined by improvements in endothelial function, systemic inflammation and cardiac and cerebral vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers (>6 months);
* Forced expiratory volume in one second/ forced vital capacity (FEV1/FVC) < 0.7 and FEV1/FVC <lower limit of normal
* Stable (>3 months exacerbation free)

Exclusion Criteria:

* On supplemental oxygen;
* Known cardiac or cerebral vascular disease, diabetes, obstructive sleep apnea;
* Uncontrolled hypertension;
* BMI >30kg/m2
* Currently performing pulmonary rehabilitation or structured exercise training;
* Desaturate during exercise (SpO2<85%)
* Cardiovascular contraindications to exercise in the incremental test used for screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | 8-weeks (following 24 sessions of exercise training)
  The change in brachial artery flow mediated dilation measured using reactive hyperaemia

SECONDARY OUTCOMES:
Arterial Stiffness | 8-weeks (following 24 sessions of exercise training)
  The change in pulse wave velocity measured using tonometry
Carotid intima-medial thickness | 8-weeks (following 24 sessions of exercise training)
  The change in carotid intima-medial thickness measured by ultrasound
Carotid Compliance | 8-weeks (following 24 sessions of exercise training)
  The change in carotid compliance measured using tonometry and ultrasound for the carotid arteries
Inflammatory Biomarkers | 8-weeks (following 24 sessions of exercise training)
  The change in serum levels of CRP, IL-6, IL-10 and TNF-alpha measured using Luminex multiplex bead-based technology
Systolic function | 8-weeks (following 24 sessions of exercise training)
  The change in stroke volume using echocardiography
Diastolic function | 8-weeks (following 24 sessions of exercise training)
  The change in left ventricular end-diastolic volume using echocardiography
Cerebral Blood Flow | 8-weeks (following 24 sessions of exercise training)
  The change in cerebral and neck blood flow using ultrasound
Cerebrovascular Reactivity | 8-weeks (following 24 sessions of exercise training)
  The change in middle cerebral artery velocity in response to carbon dioxide
Cerebrovascular Autoregulation | 8-weeks (following 24 sessions of exercise training)
  The change in phase delay measured by transfer function analysis

CONTACTS AND LOCATIONS:
Overall Officials: Neil Eves, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

REFERENCES:
- [Background] Gelinas JC, Lewis NC, Harper MI, Ainslie PN, Rolf JD, Eves ND. Aerobic Exercise Training on Peripheral Vascular Structure and Function in Patients with Chronic Obstructive Pulmonary Disease. American Journal of Respiratory and Critical Care Medicine, 191:A5305, 2015.